CLINICAL TRIAL: NCT07149415
Title: A Phase 1, Open-Label, Single-Sequence, 2-Period, Drug-Drug Interaction Study in Healthy Participants Evaluating the Effect of Omaveloxolone on the Pharmacokinetics of CYP2C19 Substrate, Omeprazole
Brief Title: A Study to Learn if Taking BIIB141 (Omaveloxolone) Affects How Omeprazole is Processed in the Body and About BIIB141's Safety in Healthy Adults Aged 18 to 55
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 296HV104
Record Dates: First submitted 2025-08-28; First posted 2025-09-02 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — omaveloxolone; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Period 1: Omeprazole (Experimental): Participants will receive a single oral dose of omeprazole on Day 1.
  Interventions: Drug: Omeprazole
- Period 2: Omaveloxolone + Omeprazole (Experimental): Participants will receive omaveloxolone from Days 2 to 15, followed by both omaveloxolone and omeprazole on Day 16.
  Interventions: Drug: Omaveloxolone; Drug: Omeprazole

INTERVENTIONS:
Drug: Omaveloxolone — Oral capsules
  Other Names: BIIB141; RTA-408
  Arms: Period 2: Omaveloxolone + Omeprazole
Drug: Omeprazole — Oral tablet

SUMMARY:
In this study, researchers will learn more about BIIB141, also known as omaveloxolone or SKYCLARYS®. This drug has been approved, or made available for doctors to prescribe, for people with Friedrich's Ataxia (FA) who are at least 16 years old. This is called a "drug-drug interaction" study. In this kind of study, researchers are looking at what happens when 2 or more medicines affect each other in the body. This could change how 1 or both of the drugs work, either making them stronger, weaker, or causing health problems.

The main goal of this study is to learn if taking BIIB141 affects how omeprazole is processed in the body. Omeprazole is a commonly used medicine to help lower the amount of acid the stomach makes.

The main question researchers want to answer in this study is :

• How does the body process omeprazole when taken with BIIB141?

Researchers will also learn more about :

* How many participants have adverse events during the study. An adverse event is a health problem that may or may not be caused by the study drug.
* How many participants have adverse reactions during the study. An adverse reaction is a health problem that may be caused by the study drug.
* If there are any changes in the participants' overall health during the study.

This study will be done as follows:

* Participants will be screened to check if they can join the study. The screening period will be up to 28 days, after which participants will check into their study research center.
* Participants will stay at the study research center for about 17 days.
* This is an "open label" study. In this kind of study, the participants, study doctor, and site staff know which study drug the participant is taking. In this study, all participants took BIIB141 and omprezole.
* Participants will take omeprazole on Day 1 and Day 16. They will also take BIIB141 once a day from Day 2 through Day 16.
* Throughout the study, researchers will take participants' blood and urine samples. Researchers will also do other tests to check the participants' overall health and will ask participants how they are feeling.
* Each participant will be in the study for up to 45 days.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the effect of omaveloxolone on the pharmacokinetics (PK) of omeprazole in healthy adult participants.

The secondary objective of this study is to assess the effect of omaveloxolone on the PK of omeprazole and to assess the safety and tolerability of a single dose administered alone and when administered concurrently with omeprazole to healthy adult participants.

ELIGIBILITY:
Key Inclusion Criteria:

* All female participants of childbearing potential must have negative results for pregnancy tests as follows:

  1. At screening, based on a serum sample obtained within 28 days prior to initial study drug administration; and
  2. Prior to dosing, based on a serum sample obtained on Study Day -1.
* Body mass index (BMI) at screening between 18 and 32 kilograms per square meter (kg/m^2), inclusive.

Key Exclusion Criteria:

* History of any clinically significant cardiac, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease, or other major disease, as determined by the Investigator.
* Clinically significant, as determined by the Investigator, 12-lead electrocardiogram (ECG) abnormalities.
* History of, or positive test result at Screening for, human immunodeficiency virus (HIV).
* History of hepatitis C infection or positive test result at Screening for hepatitis C virus antibody (HCV Ab).
* Current hepatitis B infection [defined as positive for hepatitis B surface antigen (HBsAg) and/or total anti-HBc]. Participants with immunity to hepatitis B from previous natural infection (defined as negative HBsAg, positive anti-HBc, and positive anti-HBs) or vaccination (defined as negative HBsAg, negative anti-HBc, and positive anti-HBs) are eligible to participate in the study.
* Chronic, recurrent, or serious infection (e.g., pneumonia, septicemia, and herpes simplex virus), as determined by the Investigator, within 90 days prior to Screening or between Screening and Day -1.
* Symptoms of bacterial, fungal, or viral infection (including upper respiratory tract infection) within 14 days prior to Screening or between Screening and Day -1. Participants with local fungal infection (e.g., candidiasis, tinea) are eligible to be rescreened after successful treatment of the infection.
* Prior exposure to omaveloxolone.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2025-09-02 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC0-t) of Omeprazole | Pre-dose and at multiple timepoints post-dose on Days 1, 2, 16 and 17
Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Omeprazole | Pre-dose and at multiple timepoints post-dose on Days 1, 2, 16 and 17

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Omeprazole | Pre-dose and at multiple timepoints post-dose on Days 1, 2, 16 and 17
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to end of the study (Up to Day 17)
Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities | From Day 1 up to end of the study (Up to Day 17)
Number of Participants With Change From Baseline in Clinically Relevant Abnormalities in Vital Sign Parameters | From Day 1 up to end of the study (Up to Day 17)
Number of Participants With Change From Baseline in Clinically Relevant Abnormalities in Electrocardiogram (ECG) Parameters | From Day 1 up to end of the study (Up to Day 17)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Austin Clinical Research Unit, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/